CLINICAL TRIAL: NCT02147834
Title: Effect of Ranolazine After Deferral of Percutaneous Coronary Intervention by Fractional Flow Reserve (IMWELL3)
Brief Title: Effectiveness of Ranolazine on Reducing Chest Pain in Patients With Blockage But no Stents
Acronym: IMWELL3
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to futility
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: Gilead Sciences (Industry); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201400100
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Angina
Keywords: deferred percutaneous coronary intervention; fractional flow reserve
MeSH Terms: conditions — Angina Pectoris | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine (Active Comparator): Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Interventions: Drug: Ranolazine
- Sugar pill (Placebo Comparator): Sugar pill that looks like the drug ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Sugar pill — sugar pill manufactured to mimic ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
To determine if ranolazine improves angina symptoms at 4 months compared with placebo among patients who are deferred for receiving a Percutaneous Coronary Intervention (PCI) based on the Fractional Flow Reserve (FFR) measurement.

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo-controlled, randomized, single-center (North Florida- South Georgia VA Medical Center) study. The study objective is to determine if ranolazine improves angina symptoms at 4 months compared with placebo among patients who are deferred from having a PCI based on the FFR measurement.

Baseline Procedure:

Assessments performed exclusively to determine eligibility for this study would be done only after obtaining informed consent. Assessments performed for clinical indications (not exclusively to determine study eligibility) may be used for baseline values even if the studies were done before informed consent was obtained. The assessment will include:

* Informed Consent
* Review subject eligibility criteria
* FFR value calculated at the time of cardiac catheterization
* Review previous and concomitant medications
* Frequency of symptoms and quality of life prior to study according to Seattle Angina Questionnaire (SAQ)

Screening Visit:

The assessments to determine eligibility are:

* Review of eligibility criteria
* Review of cardiac catheterization and FFR
* Review of medications taken in the past 30 days

Subjects that meet eligibility criteria will be randomized to receive either the active drug, Ranolazine or a matching placebo (non-active drug). Staff and subjects will not know if the subject will be receiving the active drug or the placebo.

Drug schedule will be as follows:

* 1st dose of one tablet (500mg) will begin the evening of Day 1
* On Days 2-7, one tablet (500mg) two times a day (12-hours apart).
* On Day 8, increase dose of study drug to two tablets (1000mg) twice a day; once in the morning and once in the evening, 12 hours apart. This dose will continue for the duration of the study. The study drug can be taken with or without food.

Telephone Follow-up:

One week phone calls will be made to determine well being, adverse events, answer questions and remind subjects to increase the study medication dose.

Two month phone calls will be made to determine well being and adverse events.

Month 4 Follow-up:

* Frequency of symptoms and quality of life according to Seattle Angina Questionnaire (SAQ)
* Assessment of well-being
* Any hospitalizations or the need for revascularization

Subjects will take the study medication for 16 weeks and will receive a phone call from the study coordinator 30 days after last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients >= 18 years of age referred for cardiac catheterization for evaluation of cardiac symptoms ( angina, fatigue, or shortness of breath)
* At least 1 indeterminate stenosis (20-80%), fractional flow reserve (FFR) >=0.8 and PCI deferred

Exclusion Criteria:

* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) during the index procedure or anticipated within the next month
* acute coronary syndrome or cardiogenic shock
* use of strong inhibitors of CTP3A (i.e. ketoconazole, itraconazole, clarithromycin,nefazodone, nelfinavir, ritonavir, indinavir and saquinavir)
* use of inducers of CYP3A (i.e. rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort)
* liver cirrhosis
* sever renal insufficience (i.e. creatinine clearance < 30mL/min/1.73 m2)
* QTc > 500 milliseconds

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Bavry, MD, MPH, Principal Investigator — North Florida/South Georgia Veterans Health System
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 subjects enrolled. First subjected enrolled 8/7/2015 and last enrolled on 11/19/2015. enrollment discontinued early by investigator due to futility.
Groups:
- Ranolazine: Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Ranolazine: Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
- Sugar Pill: Sugar pill that looks like the drug ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Sugar pill: sugar pill manufactured to mimic ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
Period: Overall Study
Arm/Group | Ranolazine | Sugar Pill
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Sugar Pill | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Seattle Angina Questionnaire Score Change From Baseline to Month 4
Description: The Seattle Angina Questionnaire is a valid and reliable instrument that measures five clinically important dimensions of health in patients with coronary artery disease (physical limitation, anginal stability, anginal frequency, treatment satisfaction, and disease perception).
Time Frame: Change in baseline to month 4
Population: The investigator ended this project early due to futility. Do data was analyzed.
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Subjective Well Being
Description: overall feeling of well being determined from rating of excellent, good, fair or poor at baseline compared to same at month 4
Time Frame: Compare from baseline to month 4
Population: The investigator ended this study early due to futility. no data was analyzed.
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Ischemia Driven Revascularization or Hospitalization
Description: frequency of the number of reported adverse events for ischemia driven revascularization or hospitalization
Time Frame: 4 month
Population: The investigator ended this study early due to futility. No data was analyzed.
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline to 4 months.
Arm/Group | Ranolazine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No